CLINICAL TRIAL: NCT01053572
Title: Evaluation of the Role of Steroids and 10% Hypertonic Sodium Chloride in Adhesiolysis in Post Lumbar Surgery Syndrome Patients: A Prospective, Randomized, Double-Blind, Equivalence, Controlled Trial of Percutaneous Lumbar Adhesiolysis
Brief Title: Role of Steroids and 10% Hypertonic Sodium Chloride in Adhesiolysis in Post Lumbar Surgery Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pain Management Center of Paducah (Other)
Responsible Party: Principal Investigator, Laxmaiah Manchikanti, MD, Medical Director, Pain Management Center of Paducah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol 23
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Low Back Pain
Keywords: Chronic low back pain; Post lumbar laminectomy syndrome; Lower extremity pain; Local anesthetic; Steroid; Percutaneous lumbar adhesiolysis
MeSH Terms: conditions — Low Back Pain | interventions — Postoperative Period

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Celestone (Active Comparator): Group I will receive adhesiolysis, local anesthetic, 10% sodium chloride solution, and non-particulate Celestone
  Interventions: Procedure: Adhesiolysis
- sodium chloride solution (Active Comparator): Group II will receive adhesiolysis, local anesthetic, 10% sodium chloride solution, and 0.9% sodium chloride solution to substitute for non-particulate Celestone
  Interventions: Procedure: Adhesiolysis
- sodium choride solution (Active Comparator): Group III will receive adhesiolysis, local anesthetic, normal sodium chloride solution instead of 10% hypertonic sodium chloride solution and non-particulate Celestone;
  Interventions: Procedure: Adhesiolysis
- Double substitutes (Active Comparator): Group IV will receive adhesiolysis, local anesthetic, and 0.9% sodium chloride solution to substitute for the 10% hypertonic sodium chloride, and 0.9% sodium chloride solution to substitute for non-particulate Celestone
  Interventions: Procedure: Adhesiolysis

INTERVENTIONS:
Procedure: Adhesiolysis — Group I will receive adhesiolysis, local anesthetic, 10% sodium chloride solution, and non-particulate Celestone
  Other Names: Adhesiolysis in post-surgery

SUMMARY:
To evaluate the effectiveness of steroids and/or 10% hypertonic sodium chloride in percutaneous adhesiolysis in managing chronic low back and/or lower extremity pain in patients with post lumbar surgery syndrome.

To evaluate and compare the adverse event profile in all groups.

DETAILED DESCRIPTION:
Recruitment is indicated in patients with chronic low back pain and lower extremity pain secondary to post lumbar laminectomy syndrome, non-responsive to conservative therapy with physical therapy, chiropractic, medical therapy, and fluoroscopically directed epidural injections.

This is a single-center, prospective, randomized, double-blind, equivalence, controlled trial performed in an interventional pain management referral center in the United States.

The study involves 240 patients studied in 4 groups with 60 patients in each group. Randomization includes sequence generation, allocation concealment, implementation, and blinding.

Data management analysis includes sample size justification of 40 patients in each group with a power of 80% and a 0.05% 2-sided significance level. Statistical methodology includes chi-squared statistics, Fisher's exact test, t-test, and paired t-test with significance evaluated at P value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

* History of lumbar surgery of at least 6 months duration in the past
* Patients over the age of 18 years
* Patients with a history of chronic function-limiting low back pain with or without lower extremity pain of at least 6 months duration (post-surgery)
* Patients who are competent to understand the study protocol and provide voluntary, written informed consent and participate in outcome measurements.

Exclusion criteria:

* Facet joints, uncontrollable as sole pain generators
* Unstable or heavy opioid use (400 mg of morphine equivalents daily)
* Uncontrolled psychiatric disorders
* Uncontrolled medical illness
* Any conditions that could interfere with the interpretation of the outcome assessments
* Pregnant or lactating women
* Patients with a history or potential for adverse reaction(s) to local anesthetic, steroids, or hypertonic sodium chloride solution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS), Oswestry Disability Index (ODI), | Outcomes are measured at baseline and at 3, 6, 12, 18, and 24 months post-treatment.
  duration of significant pain relief, opioid intake, and return to work

SECONDARY OUTCOMES:
Adverse event profile of side effects and complications. | Adverse events are measured at baseline and at 3, 6, 12, 18, and 24 months post-treatment, and at any time during the procedure or after the procedure the adverse events are suspected or expected.
  Record side effects and any complications

CONTACTS AND LOCATIONS:
Overall Officials: Laxmaiah Manchikanti, MD, Principal Investigator — PMC of Paducah
Locations (1):
- Pain Management Center of Paducah, Paducah, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No